CLINICAL TRIAL: NCT06077058
Title: Optimizing Health Promotion Strategy to Increase Quitting Preparation in Cigarette Smokers: A Pragmatic Randomized Factorial Screening Experiment
Brief Title: Quit Smoking: Optimizing Health Promotion Strategy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Health and Medical Research Fund (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: Factorial_Trial
Record Dates: First submitted 2023-09-21; First posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-09

CONDITIONS: Smoking Cessation
Keywords: Smoking Behaviors; Smoking
MeSH Terms: conditions — Smoking Cessation; Smoking | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Factorial design with four components/factors: 1) SEE versus none; 2) NRTS versus none; 3) CBIM versus none; and 4) chatbot for smoking cessation versus none, and to 2 x 2 x 2 x 2=16 trial groups. All participants will be randomly and evenly assigned to these 16 intervention groups.
  Interventions: Other: Nicotine Replace Therapy (NRT) sampling; Behavioral: Simple exercise education (SEE); Other: Chat-based instant messaging; Other: Chatbot for smoking cessation
- Control group (No Intervention): The control group will only provide simple smoking cessation advice with no intervention after recruitment

INTERVENTIONS:
Other: Nicotine Replace Therapy (NRT) sampling — The intervention involves a Zoom/WhatsApp meeting or face-to-face session with a trained counselor who introduces NRT use, possible side effects, and patch dosage based on a previous RCT guide. An online intervention pack with a pamphlet and 1-week free NRT sample (14mg or 21mg patch) is mailed to participants. After 1 week, the counselor follows up. If participants need more patches, an additional pack is mailed, and they are advised to obtain further patches from smoking cessation services or pharmacies. NRT patch users may experience skin reactions, insomnia, or vivid dreams; if severe side effects occur, they are asked to stop using NRT.
  Arms: Intervention group
Behavioral: Simple exercise education (SEE) — All participants will be given a handgrip at study enrolment. The SEE includes a Zoom/WhatsApp meeting or face-to-face session including 1) watching a 5-minute video (www.youtube.com/watch?v=mZex2Wwy3fU) showing a chair professor of public health demonstrating the 10s-E, including the simple exercises with and without handgrip. The video also encourages participants to 1) follow the exercise instructions during the video demonstration; 2) perform the exercises whenever they experience craving or an urge to smoke during the quitting process; and 3) increase their exercise frequency and intensity as much as possible, which may also increase their grip strength. Participants will also receive a leaflet with exercise instructions and motivational messages.
  Arms: Intervention group
Other: Chat-based instant messaging — Participants will receive individualized chat-based encouragement and support messages about motivation and preparation for quit attempts using WhatsApp for 8 weeks. A trained smoking cessation counsellor will have real-time (synchronous), one-to-one interaction with the participants and provide personalized motivational, behavioural support according to the participants' needs. The conversation intensity will be flexible and depends on the participant. The conversation will also be integrated with brief advice using the Behaviour Change Techniques (BCTs) (18) and the AWARD (Ask, Warn, Advise, Refer, Do-it-again) intervention model (11). The intervention protocol will be similar as that in our previous RCT on CBIM (19). For participants who receive the SEE and NRTS, the trained counsellor shall follow-up on their compliance and provide adequate advice in adhering to these interventions.
  Arms: Intervention group
Other: Chatbot for smoking cessation — The information and access to the chatbot will be introduced to participants. Through the chatbot service, participants shall access to practical information on smoking cessation 24 hours at any time, such as details on cessation services and skills for tackling cravings. By using the second-generation chatbot, participants could receive personalized risk information and recommendations for smoking cessation, as well as reach to a counsellor through WhatsApp live chat for urgently needed advice.
  Arms: Intervention group

SUMMARY:
The goal of this factorial trail is to to optimize an intervention package to enhance quit attempt preparations, quit attempts, and tobacco abstinence among smokers without a plan to quit.

The main questions it aims to answer are:

* What are the main effects of the four intervention components for increasing quit attempt preparation?
* Are there synergistic or antagonistic interactions between components?
* Does chat-based instant message or chatbot enhance the effects of nicotine replacement therapy sampling and/or simple exercise education in increasing motivation to quit?
* When participants experienced successful quitting by using the nicotine replacement therapy patch, will other tools, such as simple exercise education, chat-based instant messages, or chatbot, could help in the process and strengthen the effects of the nicotine replacement therapy patch and solve the possible problems they may encounter in using nicotine replacement therapy patch in a timely manner?

DETAILED DESCRIPTION:
1. Aims of the project This proposed project aims to optimize an intervention package to enhance quit attempt preparations, quit attempts and tobacco abstinence among smokers without a plan to quit. We expect that this study's results would demonstrate the different main effects of physical, pharmaceutical, and psychological components and their synergistic effects on smoking cessation induction. With the revealing of different effects of individual or synergistic effects of these four intervention components, including simple exercise education, NRTS, CBIM and chatbot, future smoking cessation programs may have a more precise design of using which combinations to motivate smokers. This study will also prepare for future RCTs to explore the efficacy of single or synergistically intervention components/factors for promoting smoking cessation induction. In the long run, the proportion of intervention in quit attempts and preparation to quit would increase and meet the international level and, therefore, speed up declining smoking prevalence to a single digit.
2. Study design A pilot balanced full factorial design with four components/factors: 1) SEE versus none; 2) NRTS versus none; 3) CBIM versus none; and 4) chatbot for smoking cessation versus none, and to 2 x 2 x 2 x 2=16 trial groups. All participants will be randomly and evenly assigned to these 16 intervention groups. This study protocol complies with Declaration of Helsinki and International Conference on Harmonisation Guideline for Good Clinical Practice (ICH-GCP).
3. Subjects Inclusion criteria will include 1) being a Hong Kong resident aged ≥18 years; 2) using any tobacco products every day; 3) having WhatsApp installed on their cell phone; 4) no injuries in hands and arms; 5) no medical contraindications to NRT (no severe angina, serious cardiac arrhythmias and hypertension); and 6) no plan to quit in the next 30 days. Exclusion criteria will include smokers who 1) cannot communicate in Cantonese or read Chinese; 2) currently using smoking cessation services and medication; 3) self-reported psychosis, bipolar disorder, or on psychiatric medication; and 4) pregnant smokers. As this is a pilot study to test the feasibility of conducting a full factorial design, we will recruit (10 participants x 16 groups) 160 participants to enroll in this study.
4. Recruitment strategy In the outdoor recruitment sessions, the recruitment staff will approach and distribute souvenirs or leaflets to the smokers who are smoking for 3-4 hours in the daytime. If a smoker is willing to accept them and talk to the recruitment staff, the staff will introduce the study, invite them to consent for participation, and complete a simple baseline questionnaire for further contacts and intervention delivery. Participants who complete the enrolment procedures will be offered a HKD50 shopping voucher to compensate their time spent. We will conduct 3 follow-up calls. They will be conducted after 1 week, 1 month and 3 months. In the 1 month and 3 months follow-up calls, if the participants claim s/he has already quitted smoking for equal to or more than 7 days, we will test the carbon monoxide and codinine level. Since smokers normally have higher levels of cotinine and carbon monoxide levels, we could prove if s/he quit smoking or not. We will implement carbon monoxide detector to check the carbon monoxide level, while cotinine will be used to test the cotinine level in the saliva.
5. Intervention Factor 1: Simple exercise education (SEE) All participants will be given a handgrip at study enrolment. The SEE includes a Zoom/WhatsApp meeting or face-to-face session including 1) watching a 5-minute video (www.youtube.com/watch?v=mZex2Wwy3fU) showing a chair professor of public health demonstrating the 10s-E, including the simple exercises with and without handgrip. The video also encourages participants to 1) follow the exercise instructions during the video demonstration; 2) perform the exercises whenever they experience craving or an urge to smoke during the quitting process; and 3) increase their exercise frequency and intensity as much as possible, which may also increase their grip strength. Participants will also receive a leaflet with exercise instructions and motivational messages.

   Factor 2: NRT sampling The intervention includes a Zoom/WhatsApp meeting or face-to-face session, where a trained counsellor will introduce the instruction of NRT use and possible side effects to the participant based on an intervention guide we used in the previous RCT of NRTS. The trained counsellor will suggest the NRT patch's dosage based on his/her daily cigarette consumption. If the intervention is delivered online, an intervention pack including a pamphlet and 1-week free NRT sample (patch: 14mg or 21mg) will be mailed to the participants. At 1-week after sending the NRT, the trained counsellor will follow-up with the participant. If the participant has completed all patches and willing to use more, the counsellor will mail 1 additional pack of NRT to him/her and ask him/her to obtain more from the current smoking cessation service or purchase in pharmacy. Users of NRT patch may experience skin reactions, insomnia and/or vivid dreams. If participants experience severe side effects of NRT use, the counsellor will ask them to cease use.

   Factor 3: Chat-based instant messaging Participants will receive individualized chat-based encouragement and support messages about motivation and preparation for quit attempts using WhatsApp for 8 weeks. A trained smoking cessation counsellor will have real-time (synchronous), one-to-one interaction with the participants and provide personalized motivational, behavioural support according to the participants' needs. The conversation intensity will be flexible and depend on the participant. The conversation will also be integrated with brief advice using the Behaviour Change Techniques (BCTs) (18) and the AWARD (Ask, Warn, Advise, Refer, Do-it-again) intervention model (11). The intervention protocol will be similar as that in our previous RCT on CBIM (19). For participants who receive the SEE and NRTS, the trained counsellor shall follow-up on their compliance and provide adequate advice in adhering to these interventions.

   Factor 4: Chatbot for smoking cessation The information and access to the chatbot will be introduced to participants. Through the chatbot service, participants shall access to practical information on smoking cessation 24 hours at any time, such as details on cessation services and skills for tackling cravings. By using the second-generation chatbot, participants could receive personalized risk information and recommendations for smoking cessation, as well as reach to a counsellor through WhatsApp live chat for urgently needed advice.
6. Randomization, allocation concealment and blinding The random allocation sequence will be computer-generated by an investigator who has no other involvement in the study. Simple individual randomization by sequentially numbered, opaque sealed envelopes (SNOSE) will be used to ensure the recruitment staff and the participants will be concealed in the allocation sequence before the group allocation.

   Blinding of participants and the research staff who deliver the intervention will not be possible. Follow-up outcome assessments will be conducted by research assistants who will be blinded for the group allocation.
7. Evaluation plan To examine whether the intervention can be delivered as it is designed (scalability), we will evaluate the intervention fidelity and smokers' adherence to the intervention. Regarding to SEE, counsellors will document the time spent on delivering the SEE and participants' response. Regarding NRTS, counsellors will document the time spent on medication advice, what will be included in the advice, and any side effects or concerns reported by the participants at 1-week follow-up. Regarding CBIM, number of messages sent by counsellors and the participants will be documented. For chatbot, number of messages sent by participants will be recorded.
8. Data analyses All statistical analysis will be conducted in STATA/MP version 16.1. The primary analysis will examine the intervention's main and interaction effects on the primary outcome by intention-to-treat, assuming non-respondents at follow-up are smokers without quit attempts. Between-subject factorial linear mixed model (LMM) will be used to evaluate the main effects, six 2-way interactions (SEE X NRTS, SEE X CBIM, NRTS X CBIM, SEE X chatbot, NRTS X chatbot, CBIM X chatbot), four 3-way interaction (SEE X NRT X CBIM, SEE X NRT X chatbot, SEE X CBIM X chatbot and NRT X CBIM X chatbot) and one 4-way interaction (SEE X NRTS X CBIM x chatbot) using effect coding (levels are coded -1 and +1) on IBC-S. Analyses will be adjusted for demographics and smoking-related covariates, and supplemented with multiple imputation and complete-case analysis. The IBC-S score of sub-groups involved in a significant interaction (5% level of significance) will be plotted on a bar chart to visualize the comparisons.
9. Direct access to source data/documents The raw data will be stored in the CD-ROM and locked in a cupboard with keys kept by the Principal Investigator. Only the Investigators and Research Assistants of the project will be permitted access to raw data and/or study records. The data will be kept for 10 years after the study is completed.
10. Dissemination of study result The initial findings will be submitted for application for the coming round of the Health Medical Research Fund or the General Research Fund. The findings will be disseminated through publication in the journal Addiction or other peer-reviewed journals. Also, the findings will be useful evidence for expert comments or deputations of smoking-related issues in the Legislation Council.
11. Consent Eligible participants will be invited to participate in the study by obtaining written consent.

ELIGIBILITY:
Inclusion Criteria:

* Being a Hong Kong resident aged ≥18 years;
* Using any tobacco products every day;
* Having WhatsApp installed on their cell phone;
* No injuries in hands and arms;
* No medical contraindications to NRT (no severe angina, serious cardiac arrhythmias and hypertension); and
* No plan to quit in the next 30 days.

Exclusion Criteria:

* Cannot communicate in Cantonese or read Chinese;
* Currently using smoking cessation services and medication;
* Self-reported psychosis, bipolar disorder, or on psychiatric medication; and
* Pregnant smokers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Incremental Behaviour Change toward Smoking cessation (IBC-S) | 3-month
  This 15-item scale measures a spectrum of behaviours and cognitions antecedent to prepare smoking cessation. The minimum value is 3 and the maximum value is 27. Higher scores mean a better outcome.

SECONDARY OUTCOMES:
The proportion of smokers who self report quit attempts | 3-month
Self-reported tobacco abstinence in the past 30 days | 3-month
Biochemically validated abstinence | 3-month
Time spend for offering simple exercise education (SEE) | Baseline
  Counsellors will document the time spent on delivering the SEE and participants' response.
Time spent on Nicotine Replacement Therapy (NRT) medication advice | Baseline
  Counsellors will document the time spent on medication advice
Number of chatbased instant messages (CBIM) sent by counsellors and the participants | 3-month
  Number of messages sent by counsellors and the participants will be documented
Number of Chatbot messages sent by participants | 3-month
The time interval between getting smokers contact information and initiate conversation with smokers | 3-month
Percentage of smokers CBIM offers social support of smoking cessation induction | 3-month
  <25% of the conversation; 25%-75% of the conversation; >75% of the conversation
Percentage of CBIM counselor messages reply to smokers questions within 2 hours | 3-month
  <25% of the time; 25%-75% of the time; >75% of the time
Percentage of CBIM smokers reply to a counselor when necessary | 3-month
  <25% of the time; 25%-75% of the time; >75% of the time
Percentage of CBIM counselor communicates with smokers in a respectful, positive, and non-judgmental manner | 3-month
  <25% of the time; 25%-75% of the time; >75% of the time
Percentage of counselor follows counseling guideline | 3-month
  <25% of the conversation; 25%-75% of the conversation; >75% of the conversation
Percentage of counselor uses behavior change technique during the conversation for coping with smoking | 3-month
  <25% of the conversation; 25%-75% of the conversation; >75% of the conversation
Percentage of counselor reminds smokers to practice brief exercise | 3-month
  <25% of the conversation; 25%-75% of the conversation; >75% of the conversation
Percentage of counselor remind smokers to use NRT sample | 3-month
  <25% of the conversation; 25%-75% of the conversation; >75% of the conversation
Percentage of smokers replied doing exercise after reminding | 3-month
  <25% of the conversation; 25%-75% of the conversation; >75% of the conversation
Percentage of smokers replies using NRT after reminding | 3-month
  <25% of the conversation; 25%-75% of the conversation; >75% of the conversation
Number of handgrip delivered by counselor | Baseline
Number of handgrip received by smokers | Baseline
Time spend of watching SEE video | Baseline
Number of smokers attend simple exercise education session | Baseline
Time spend of smokers watching video | Baseline
Number of smokers practice exercise after watching video | 3-month
Number of NRT sample prescribe by counselor | Baseline
Number of NRT sample receive by smokers | Baseline
Number of NRT sample used (Dose (Days used and patches used)) | Baseline
Numbe of smokers purchase NRT after used up NRT sample over-the-counter | Baseline
Number of smokers request NRT full-package from TWGHs after used NRT sample | Baseline
Number of smokers use NRT after used up NRT sample | Baseline
Percentage of counselor introduce places where smokers can get NRT | Baseline
  <25% of the conversation; 25%-75% of the conversation; >75% of the conversation
Percentage of counselor introduce reasons for using NRT sample | Baseline
  <25% of the conversation; 25%-75% of the conversation; >75% of the conversation
Percentage of counselor introduce withdrawal symptoms of smoking cessation | Baseline
  <25% of the conversation; 25%-75% of the conversation; >75% of the conversation
Percentage of counselor Introduce how to use NRT sample and tips | Baseline
  <25% of the conversation; 25%-75% of the conversation; >75% of the conversation
Percentage of counselor introduce possible adverse effects of NRT sample | Baseline
  <25% of the conversation; 25%-75% of the conversation; >75% of the conversation
Percenage of counselor offer other suggestions of smoking cessation (e.g., tell your family member that you are using NRT, practice various exercise and keep a healthy diet in case of weight gain during smoking cessation) | Baseline
  <25% of the conversation; 25%-75% of the conversation; >75% of the conversation
Percenage of counselor refer smokers to other smoking cessation agencies | 3-month
  <25% of the conversation; 25%-75% of the conversation; >75% of the conversation
Number of smokers agree to referral | 3-month

OTHER OUTCOMES:
Covariate 1 | Baseline
  Age (Target range should be above 18 years old)
Covariate 2 | Baseline
  Gender (Female/Male)
Covariate 3 | Baseline
  Martial Status (Response: Single/ Married/ Divorced/ Widowed)
Covariate 4 | Baseline
  Monthly household income (Response: HK$5,999 and below, HK$6,000-9,999, HK$10,000-19,999, HK$20,000-29,999, HK$30,000-39,999, HK$40,000-59,999, HK$60,000 and above, no income, not clear/difficult to answer, refuse to answer).
Covariate 5 | Baseline
  Employment status (Response: Student/ Self-employed/ Employed/ Unemployed/ Full time taking care family/ Retired)
Covariate 6 | Baseline
  Job nature (Response: Management/ Professional/ Professional Assistant/ Clerk/ Service-related and sales/ Fisheries and Agriculture workers/ handicraft-related/ machine controlled-related/ non-worker/ Refuse to answer/ Difficult to classified)
Covariate 7 | Baseline
  Highest Educational level (Reponse: Primary school or below/ Junior high school/ high school/ bachlor degree or above)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Research data and documentation will be available upon request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 3 years after the completion of the relevant publications

REFERENCES:
- [Result] Census & Statistics Department (Hong Kong SAR government. In: Thematic Household Survey, Report No 70: Pattern of Smoking. Hong Kong: Census & Statistics Department; 2020.
- [Result] Leung DY, Chan SS, Chan V, Lam TH. Hardcore smoking after comprehensive smoke-free legislation and health warnings on cigarette packets in Hong Kong. Public Health. 2016 Mar;132:50-6. doi: 10.1016/j.puhe.2015.10.007. Epub 2015 Nov 21. PMID 26612457
- [Result] Richter KP, Ellerbeck EF. It's time to change the default for tobacco treatment. Addiction. 2015 Mar;110(3):381-6. doi: 10.1111/add.12734. Epub 2014 Oct 16. PMID 25323093
- [Result] Flocke SA, Step MM, Lawson PJ, Smith S, Zyzanski SJ. Development of a Measure of Incremental Behavior Change Toward Smoking Cessation. Nicotine Tob Res. 2017 Dec 13;20(1):73-80. doi: 10.1093/ntr/ntw217. PMID 27613910
- [Result] Ali A, Kaplan CM, Derefinko KJ, Klesges RC. Smoking Cessation for Smokers Not Ready to Quit: Meta-analysis and Cost-effectiveness Analysis. Am J Prev Med. 2018 Aug;55(2):253-262. doi: 10.1016/j.amepre.2018.04.021. Epub 2018 Jun 12. PMID 29903568
- [Result] Catley D, Goggin K, Harris KJ, Richter KP, Williams K, Patten C, Resnicow K, Ellerbeck EF, Bradley-Ewing A, Lee HS, Moreno JL, Grobe JE. A Randomized Trial of Motivational Interviewing: Cessation Induction Among Smokers With Low Desire to Quit. Am J Prev Med. 2016 May;50(5):573-583. doi: 10.1016/j.amepre.2015.10.013. Epub 2015 Dec 23. PMID 26711164
- [Result] Carpenter MJ, Hughes JR, Gray KM, Wahlquist AE, Saladin ME, Alberg AJ. Nicotine therapy sampling to induce quit attempts among smokers unmotivated to quit: a randomized clinical trial. Arch Intern Med. 2011 Nov 28;171(21):1901-7. doi: 10.1001/archinternmed.2011.492. PMID 22123796
- [Result] Amante DJ, Blok AC, Nagawa CS, Wijesundara JG, Allison JJ, Person SD, Morley J, Conigliaro J, Mattocks KM, Garber L, Houston TK, Sadasivam RS. The 'Take a Break' game: Randomized trial protocol for a technology-assisted brief abstinence experience designed to engage lower-motivated smokers. Contemp Clin Trials. 2020 Jun;93:106002. doi: 10.1016/j.cct.2020.106002. Epub 2020 Apr 23. PMID 32335288
- [Result] Chan SS, Wong DC, Cheung YT, Leung DY, Lau L, Lai V, Lam TH. A block randomized controlled trial of a brief smoking cessation counselling and advice through short message service on participants who joined the Quit to Win Contest in Hong Kong. Health Educ Res. 2015 Aug;30(4):609-21. doi: 10.1093/her/cyv023. Epub 2015 Jun 25. PMID 26116584
- [Result] Cheung YTD, Chan CHH, Ho KS, Tang C, Lau CWH, Li WHC, Wang MP, Lam TH. Effectiveness of nicotine replacement therapy sample at outdoor smoking hotspots for initiating quit attempts and use of smoking cessation services: a protocol for a cluster randomised controlled trial. BMJ Open. 2020 Apr 7;10(4):e036339. doi: 10.1136/bmjopen-2019-036339. PMID 32269028
- [Result] Collins LM. Optimization of Behavioral, Biobehavioral, and Biomedical Interventions: The Multiphase Optimization Strategy (MOST) [Internet]. Cham: Springer International Publishing; 2018 [cited 2021 Feb 9]. (Statistics for Social and Behavioral Sciences). Available from: http://link.springer.com/10.1007/978-3-319-72206-1
- [Result] Cheung YTD, Cheung Li WH, Wang MP, Lam TH. Delivery of a Nicotine Replacement Therapy Sample at Outdoor Smoking Hotspots for Promoting Quit Attempts: A Pilot Randomized Controlled Trial. Nicotine Tob Res. 2020 Aug 24;22(9):1468-1475. doi: 10.1093/ntr/ntz138. PMID 31404466
- [Result] Wang MP, Luk TT, Wu Y, Li WH, Cheung DY, Kwong AC, Lai V, Chan SS, Lam TH. Chat-based instant messaging support integrated with brief interventions for smoking cessation: a community-based, pragmatic, cluster-randomised controlled trial. Lancet Digit Health. 2019 Aug;1(4):e183-e192. doi: 10.1016/S2589-7500(19)30082-2. Epub 2019 Jul 31. PMID 33323188
- [Result] Weng X, Luk TT, Suen YN, Wu Y, Li HCW, Cheung YTD, Kwong ACS, Lai VWY, Chan SSC, Lam TH, Wang MP. Effects of simple active referrals of different intensities on smoking abstinence and smoking cessation services attendance: a cluster-randomized clinical trial. Addiction. 2020 Oct;115(10):1902-1912. doi: 10.1111/add.15029. Epub 2020 Mar 25. PMID 32149425
- [Result] Cheung YT, Lam TH, Chan CHH, Ho KS, Fok WYP, Wang MP, Li WHC. Brief handgrip and isometric exercise intervention for smoking cessation: A pilot randomized trial. Addict Behav. 2020 Jan;100:106119. doi: 10.1016/j.addbeh.2019.106119. Epub 2019 Sep 4. PMID 31522134
- [Result] Fiore MC, Jaén CR, Baker TB, Bailey WC, Benowitz NL, Curry SJ. Treating tobacco use and dependence: 2008 update-clinical practice guideline. 2008. Rockville, MD: Public Health Service, US Department of Health and Human Services; 2008.
- [Result] Cheung YTD, Lam TH, Li WHC, Wang MP, Chan SSC. Feasibility, Efficacy, and Cost Analysis of Promoting Smoking Cessation at Outdoor Smoking "Hotspots": A Pre-Post Study. Nicotine Tob Res. 2018 Nov 15;20(12):1519-1524. doi: 10.1093/ntr/ntx147. PMID 28655173
- [Result] Michie S, Hyder N, Walia A, West R. Development of a taxonomy of behaviour change techniques used in individual behavioural support for smoking cessation. Addict Behav. 2011 Apr;36(4):315-9. doi: 10.1016/j.addbeh.2010.11.016. Epub 2010 Dec 15. PMID 21215528
- [Result] Luk TT, Wong SW, Lee JJ, Chan SS, Lam TH, Wang MP. Exploring Community Smokers' Perspectives for Developing a Chat-Based Smoking Cessation Intervention Delivered Through Mobile Instant Messaging: Qualitative Study. JMIR Mhealth Uhealth. 2019 Jan 31;7(1):e11954. doi: 10.2196/11954. PMID 30702431